CLINICAL TRIAL: NCT02347397
Title: A Prospective, Randomized, Multicenter Clinical Study in Elderly Chinese Subjects to Compare the Safety and Efficacy of the SS Bipolar Head and SL-TWIN Stem With Bipolar Head and SL-PLUS Stem in Hemiarthroplasty of the Hip
Brief Title: Project JAY HAP Registration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew Orthopaedics (Beijing) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-4561-01
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SS Bipolar Head + SL-TWIN Stem (Experimental): Subject will be implanted with the SS Bipolar Head & SL-TWIN Stem
  Interventions: Device: SS Bipolar Head + SL-TWIN Stem
- Bipolar Head + SL-PLUS Stem (Active Comparator): Subject will be implanted with the Bipolar Head & SL-PLUS Stem
  Interventions: Device: Bipolar Head + SL-PLUS Stem

INTERVENTIONS:
Device: SS Bipolar Head + SL-TWIN Stem — Subject will undergo hemiarthroplasty surgery with SS Bipolar Head & SL-TWIN Stem
  Arms: SS Bipolar Head + SL-TWIN Stem
Device: Bipolar Head + SL-PLUS Stem — Subject will undergo hemiarthroplasty surgery with Bipolar Head & SL-PLUS Stem
  Arms: Bipolar Head + SL-PLUS Stem

SUMMARY:
This is a prospective, randomized, multicenter clinical study in elderly Chinese subjects to compare the safety and efficacy of the SS Bipolar Head and SL-TWIN Stem with Bipolar Head and SL-PLUS Stem in hemiarthroplasty of the hip

DETAILED DESCRIPTION:
Elderly patients, especially post-menopausal women, often suffer a femoral neck fracture due to osteoporosis, even with very little trauma. Femoral neck fracture is a common disease in elderly patients, it accounts for 3.6% of total body fractures. In China, as the population continues to age and life expectancy increases, the incidence of femoral neck fracture has significantly increased.

Hip replacement surgery includes total hip arthroplasty (THA) and hemiarthroplasty (HAP). Hemiarthroplasty of the hip involves replacement of the diseased, affected, or broken femoral head and/or neck with a prosthetic component. Hemiarthroplasty does not involve resurfacing of the acetabulum, and therefore a bipolar or unipolar prosthetic head articulates against the host acetabular articular cartilage. Avoiding the need, when appropriate, to resurface the acetabulum helps to minimize surgical trauma, operative time and dislocation risk, while preserving acetabular bone stock. These also result in shorter bed stay and faster recovery comparing with the THA.

There has been an increase in imported hip prostheses during the past decade, so that surgeons now have more choices of implants. However, the high cost of imported prostheses has become a barrier to the development of hip replacement in China and caused many patients requiring immediate hip replacement to have to delay or miss their surgery. The development and promotion of high-quality domestic joint implants and surgical instruments is the key to the development of joint replacement technique in China.

The primary objective of this study is to demonstrate non-inferiority of subjects implanted with the SS Bipolar Head + SL-TWIN Stem compared to a randomized concurrent control group of subjects implanted with the Bipolar Head + SL-PLUS Stem in terms of mean Harris Hip Score (HHS) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 65 and 90 years inclusive of Chinese ethnicity.
* Subject presents with femoral neck fracture (Garden Type II, III, or IV) requiring hemiarthroplasty of the hip.
* Subject is able to move independently before the fracture, with or without the use of walking aids .
* Subject who is able to give voluntary, written informed consent to participate in the study and from whom consent has been obtained by signing and dating an EC-approved consent form.
* Subject who is able to understand this clinical study, co-operates with the investigational procedures and is willing to return to the hospital for all the required post-operative follow-ups for up to 12 months.
* Life expectancy of subject is over 2 years.

Exclusion Criteria:

* Bilateral hip disease with the anticipated need for bilateral hip implant during study participation (i.e., within the next 12 months).
* Subject experienced prior joint replacement surgery on any major joint (hip, knee) in lower limb within the last 12 months.
* Subject has known or suspected metal sensitivity.
* Subject is known to have insufficient bone stock resulting from conditions such as cancer, significant osteoporosis or metabolic bone disorders, which cannot provide adequate support and/or fixation to the prosthesis.
* Subject is severely obese (BMI>35).
* Subject is not suitable for hemiarthroplasty (i.e., inflammatory arthritis, pathological fractures, etc.)
* Subject had an active infection or sepsis (treated or untreated)
* Subject has conditions that may compromise implant stability or postoperative recovery (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency, hip abduction muscle strength less than grade IV or complete loss, or neuromuscular disease).
* Subject has an emotional or neurological condition that would affect their ability or willingness to participate in the study (e.g. cognitive disorder, mental illness, mental retardation).
* Subject is immunosuppressed, has an autoimmune disorder, or an immunosuppressive disorder. For examples, subject is on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses) or has acquired immunodeficiency syndrome (AIDS).
* Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.
* Subject was enrolled in another investigational drug, biologic, or device study in the last 12 months.
* Known alcohol and/or drug abuse

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 1 year post-operative

SECONDARY OUTCOMES:
Composite Clinical Success, as indicated by A) No revision of any device component; and B) Total Harris Hip Score greater than or equal to 80 (excellent to good score); and C) Radiologic success. | 1 year post-operative
  A successful individual outcome for a subject in hemiarthroplasty will be characterized at 1 year postoperative by a composite of three success criteria:
  A. No revision of any device component; and B. Total Harris Hip Score greater than or equal to 80 (excellent to good score); and C. Radiologic success.

OTHER OUTCOMES:
Barthel Index | 1 year post-operative
SF-12 Health Survey | 1 year post-operative
Number of adverse events | Up to 1 year post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (5):
- China (5):
  - Haikou People's Hospital, Haikou, Hainan
  - Luoyang Orthopedic-Traumatological Hospital, Luoyang, Henan
  - Inner Mongolia Bao Gang Hospital, Baotou, Inner Mongolia
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No